CLINICAL TRIAL: NCT03166163
Title: Evaluation of Bleeding on Brushing Among a Group of Egyptian Children After Using Azadirachta Indica (Neem Extract)Mouthwash Versus Chlorhexidine Mouthwash: A Randomized Controlled Trial
Brief Title: Evaluation of Bleeding on Brushing Using Neem Extract Mouthwash Versus Chlorhexidine Mouthwash
Acronym: mouthwash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Sherif Ali Mostafa, Master dental student, pediatric dentistry department., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2621985; 2621985 (Other: CairoU)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Gingival Bleeding
Keywords: bleeding on brushing
MeSH Terms: conditions — Gingival Hemorrhage | interventions — neem oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This was a double -blind study as the investigator was unaware about the sampling of the groups and study subjects were unaware about the mouthwash they were using
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azadirachta indica (Neem extract) (Experimental): its herbal mouthwash that will be given to a group a Egyptian children twice a day(10 ml each) for 3 weeks
  Interventions: Drug: Azadirachta indica
- chlorhexidine mouthwash (Active Comparator): its an antimoicrobial, antiplaque mouthwash that will be given to a group of Egyptian children twice daily(10 ml each) for 3 weeks
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Azadirachta indica — Its a herbal mouthwash that will be given to group of Egyptian Children twice daily for 3 weeks
  Other Names: neem extract
  Arms: Azadirachta indica (Neem extract)
Drug: Chlorhexidine mouthwash — its an antimocrobial, antiplaque mouthwash that will be given to a group of Egyptian children twice daily (10 ml each) for 3 weeks
  Other Names: chlohexidine
  Arms: chlorhexidine mouthwash

SUMMARY:
i will compare the effect of neem extract mouthwash versus the chlorhexidine mouthwash on bleeding on brushing among a group of Egyptian children.

DETAILED DESCRIPTION:
1. First , we will select the patients according to the inclusion criteria.
2. We will take sulcus bleeding index which is defined as an index of gingival inflammation in which bleeding is measured from four gingival units using a periodontal probe. The scoring is ranging around eight anterior teeth from 0 to 5.In this study, we will take only score 2 which is bleeding on probing, change in colour and no edema in order to reduce variability.
3. 2%neem extract will be used to prepare mouthwash while, chlorhexidine will be used as positive control.
4. Chlorhexidine will be coded with the letter "A" and the mouthwash of 2%neem extract with the letter "B".
5. The participants included will be allocated into 2 groups by drawing of sealed and opaque envelopes containing the codes "A" and "B"
6. The intra and extraoral examinations will be made using masks, gloves, cap, goggles, gauze, medical tray, dental mirror and WHO probe. All materials will be packaged in sterilization wraps and autoclaved, following the required biosafety standards.
7. The rinses will be performed twice daily, which will be supervised by the parents legal guardians previously instructed. Kits containing toothpaste an brush will be provided, so that the patients will use the same toothpaste, avoiding any interference with the results.
8. After 3 weeks, we will ask the patient if there is any gingival bleeding in addition we will measure the sulcus bleeding index.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children aged 8-10 years old with gingivitis

  2. cooperative children

  3.both genders

  4.medically free

  5. sulcus bleeding index score is 2

Exclusion Criteria:

* 1. Children undergoing orthodontic treatment

  2.Children undergoing any other oral hygiene aid other than routine teeth brushing

  3.Children with known history of allergy to any mouthwash or drug

  4.Parents unable to give informed consent

  5.Children taking antibiotic or antiseptic in previous two months

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-06-11 (Estimated); Study Completion 2017-06-11 (Estimated)

PRIMARY OUTCOMES:
Bleeding on brushing | 3 weeks
  measuring device(asking the patient) measuring unit (binary)

SECONDARY OUTCOMES:
sulcus bleeding index | 3 weeks
  measuring device (measuring the sulcus bleeding index) measuring unit (the score of the sulcus bleeding index)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B Eltaweel, Ass. prof, Study Director — Cairo University
Locations (1):
- Samar Sherif Ali Moustafa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
it will be available when it is finished

REFERENCES:
- [Background] Balappanavar AY, Sardana V, Singh M. Comparison of the effectiveness of 0.5% tea, 2% neem and 0.2% chlorhexidine mouthwashes on oral health: a randomized control trial. Indian J Dent Res. 2013 Jan-Feb;24(1):26-34. doi: 10.4103/0970-9290.114933. PMID 23852229
- [Background] Dhingra K, Vandana KL. Effectiveness of Azadirachta indica (neem) mouthrinse in plaque and gingivitis control: a systematic review. Int J Dent Hyg. 2017 Feb;15(1):4-15. doi: 10.1111/idh.12191. Epub 2016 Feb 15. PMID 26876277
- See also: Comparison of the effectiveness of 0.5% tea, 2% neem and 0.2% chlorhexidine mouthwashes on oral health: a randomized control trial. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Comparison+of+the+effectiveness+of+0.5%25+tea%2C+2%25+neem+and+0.2%25+chlorhexidine+mouthwashes+on+oral+health%3A+a+randomized+control+trial.
- See also: Effectiveness of Azadirachta indica (neem) mouthrinse in plaque and gingivitis control: a systematic review. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Effectiveness+of+Azadirachta+Indica+(neem)+mouthrinse+in+plaque+and+gingivitis+control%3Aa+systematic+review